CLINICAL TRIAL: NCT02905981
Title: Triferic (Ferric Pyrophosphate Citrate) Administered Orally With Shohl's Solution for the Treatment of Iron-Refractory Iron-Deficiency Anemia
Brief Title: Triferic IRIDA (Iron-Refractory Iron-Deficiency Anemia) Protocol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited subjects, patient compliance
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-15
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Iron-Refractory Iron-Deficiency Anemia
Keywords: IRIDA; Triferic; soluble ferric pyrophosphate; Shohl's solution
MeSH Terms: conditions — Iron-Refractory Iron Deficiency Anemia | interventions — ferrous sulfate; Citrates; Citric Acid; ferric pyrophosphate; spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Period 1: Iron Absorption Tests (Experimental): During 3 consecutive weekly study visits, patients will receive Fer-In- Sol orally 3 milligram iron per kilogram (mg Fe/kg) body weight, Shohl's solution 0.67 millimoles per kilogram (mmol/kg) followed 5 - 15 minutes later by Fer-In- Sol orally 3 mg Fe/kg body weight, and Shohl's solution 0.67 mmol/kg followed 5 - 15 minutes later by Triferic orally 3 mg Fe/kg body weight (respectively). All oral doses will be administered by study personnel at the research center. Blood tests will be conducted following each administration in order to measure iron absorption to see if patients qualify for Period 2.
  Interventions: Drug: Fer-In-Sol; Drug: Shohl's solution; Drug: Triferic
- Period 2: Dose Titration (Experimental): Patients who qualified as 'Triferic responders' in Period 1 will participate in Period 2. Patients will be given oral Shohl's solution and Triferic to administer at home 3 times per day, with the dose being titrated higher or lower based on lab results. The initial dose will be the same as Period 1 (Shohl's solution 0.67 mmol/kg followed 5 - 15 minutes later by Triferic orally 3 mg Fe/kg body weight) but may be adjusted during Period 2 based on lab results. Period 2 will involve 5 study visits, scheduled every 4 weeks. At the end of Period 2, blood tests will be performed to determine if patients qualify for Period 3.
  Interventions: Drug: Shohl's solution; Drug: Triferic
- Period 3: Hemoglobin Maintenance (Experimental): Patients who qualified as 'hemoglobin responders' in Period 2 will participate in Period 3. Patients will continue to take Shohl's solution and Triferic at their titrated dose for an additional six months to confirm that their hemoglobin can be maintained over an extended period of time. The period will be comprised of 3 study visits, scheduled every 8 weeks.
  Interventions: Drug: Shohl's solution; Drug: Triferic

INTERVENTIONS:
Drug: Fer-In-Sol — Fer-In-Sol is an over-the-counter oral iron supplement. It will be administered during Period 1 at a dose of 3 mg/kg body weight.
  Other Names: FeSO4
  Arms: Period 1: Iron Absorption Tests
Drug: Shohl's solution — Shohl's solution will be supplied as 500-milliliter (mL) bottles containing citric acid United States Pharmacopeia (USP) 640 milligrams per 5 milliliters (mg/5 mL) and hydrous sodium citrate USP 490 mg/5 mL. It will be administered during all Periods at a dose of 0.67 mmol/kg body weight.
  Other Names: Citrate; Oracit
Drug: Triferic — Triferic is an iron salt that is approved by the Food and Drug Administration (FDA) for the maintenance of hemoglobin in patients with end stage kidney disease on hemodialysis. It is experimental in this study because it has not yet been approved for patients with IRIDA. It will be administered during Period 1 at a dose of 3 mg/kg body weight. In Periods 2 and 3 the dose may be adjusted based on lab results.
  Other Names: ferric pyrophosphate citrate (FPC)

SUMMARY:
The main purpose is to determine whether Triferic, administered orally with Shohl's solution, is safe and effective for the treatment of iron-refractory iron-deficiency anemia (IRIDA).

DETAILED DESCRIPTION:
This is an open label, 3-period study assessing the safety, efficacy, and pharmacokinetics of Triferic and Shohl's solution administered orally to patients with IRIDA. A total of 28 patients stratified by 4 age groups (age 0 to <6 years, age 6 to <12 years, age 12 to <18 years, and age >=18 years) will be studied.

Total participation in the study is between 4 weeks (Period 1) and 12 months (Periods 1, 2, and 3), depending upon how many Periods each patient participates in. Following screening, in Period 1 (iron absorption testing) patients undergo oral iron absorption testing during 3 visits to confirm that they adequately absorb iron from Triferic when it is administered with Shohl's solution ('Triferic responders': patients with a maximal increase from baseline in serum iron concentration >100 micrograms per deciliter (μg/dL) following an oral Shohl's solution and Triferic dose).

The 'Triferic responders' from Period 1 are then invited to participate in Period 2 (dose titration). The patients will receive Shohl's solution and Triferic orally up to 3 times per day for 4 months, titrated as needed based on laboratory results and patient tolerance, to determine whether their hemoglobin levels respond to this treatment. Period 2 'hemoglobin responders' (patients with an increase from baseline in hemoglobin (Hgb) concentration ≥1.0 grams per deciliter (g/dL) at Visit 9) will be invited to participate in period 3.

In Period 3 patients will receive Shohl's solution and Triferic orally up to 3 times per day for an additional 6 months to determine whether the hemoglobin response observed in Period 2 is sustainable. During Period 3, Shohl's solution and Triferic dose and frequency may continue to be titrated as needed based on laboratory results and patient tolerance.

A follow-up visit will occur approximately 1 week after the last completed Period study visit, regardless of the Period that the patient completes the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients have provided informed consent and have signed the informed consent form. For pediatric patients, parents/legal guardians of the patient have the ability to understand the requirements of the study and have demonstrated a willingness to have their child comply with all study procedures by signing the informed consent form. Where applicable, assent of the pediatric patient has also been obtained for all study procedures prior to any study-related activities.
2. Patient has a history of congenital hypochromic microcytic anemia.
3. Patient has a mean corpuscular volume (MCV) ≤75 fluid ounce (fL) at screening.
4. Patient has a serum transferrin saturation ≤15% at screening.
5. Patient has a history of no or incomplete response to oral iron therapy.
6. Patient has a history of no or incomplete response to intravenous iron administration.
7. Patient has a history of hepcidin concentration ≥10 nanograms per milliliter (ng/mL) (3.58 nanometer (nM)) off iron supplements, adjusted for the specific hepcidin assay used to be at least 1 standard deviation (SD) greater than the mean for patients with iron-deficiency anemia.
8. Patient is documented to have homozygous or compound heterozygous pathogenic mutations in Transmembrane Serine Protease 6 (TMPRSS6) in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
9. Patient has appropriate laboratory values for their disease state at screening (per investigator judgment).
10. Patient has no significant abnormal findings on physical examination at screening that would preclude participation in the study (per investigator judgment).
11. If the patient is female, she must be pre-pubertal, have had documented surgical sterilization ≥2 years prior to screening, or be practicing adequate birth control. All female patients 9 years of age and older, and also any who have reached menarche before age 9 years, must have a negative serum pregnancy test during screening. It is the investigator's responsibility to determine whether the patient has adequate birth control for study participation.

Exclusion Criteria:

1. Patient has had intravenous (IV) or oral iron supplements within 2 weeks prior to Visit 2.
2. Patient has had a blood transfusion within 3 months prior to Visit 2.
3. Patient is receiving intravenous or oral antibiotics or antifungals for any infectious process. Prophylactic antibiotics administered on a regular basis are allowed. Otherwise-eligible patients may be rescreened when they have recovered from any acute illnesses.
4. Patient has a body weight of <11 lbs (5 kg) at screening.
5. Patient has participated in an investigational drug study within the 30 days prior to Visit 2.
6. Patient has any condition that, in the opinion of the investigator, is likely to prevent the patient from complying with or successfully completing the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01-17; Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD, FACP, Study Director — Rockwell Medical, Inc

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: In this phase 2, open-label, 3-period study all participants enrolled underwent an oral iron absorption testing with Triferic when it is administered with Shohl's solution during 3 visits during Period 1. In Period 2 (dose titration), the patients received Shohl's solution and Triferic orally up to 3 times per day for 4 months. In Period 3 patients received Shohl's solution and Triferic orally up to 3 times per day for an additional 6 months
Period: Overall Study
Arm/Group | All Participants
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- All Patients in Study: All patients enrolled in the study who undergoing all three periods: an oral iron absorption testing period (Period 1), a Triferic dose titration period (Period 2), a hemoglobin maintenance period (Period 3
Arm/Group | All Patients in Study
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of Triferic Delivered to IRIDA Patients:Change in Hemoglobin (Hgb)
Description: The efficacy will be done by assessing the change from baseline in hemoglobin concentration
Time Frame: 4 months
Measure: Number; unit: micrograms per deciliter
Arm/Group | All Patients in Study
Number analyzed (Participants) | 1
micrograms per deciliter | 7.9

2. Secondary Outcome: The Efficacy of Triferic Being Delivered to Iron-refractory Iron Deficiency Anemia (IRIDA) Patients:Change in Serum Iron
Description: The efficacy will be done by assessing the change from baseline in serum iron
Time Frame: 4 months
Measure: Number; unit: micrograms per deciliter
Arm/Group | All Patients in Study
Number analyzed (Participants) | 1
micrograms per deciliter | 19

3. Secondary Outcome: The Efficacy of Triferic Being Delivered to IRIDA Patients:Change From Baseline in Transferrin Saturation (TSAT)
Description: The efficacy will be done by assessing the change from baseline in TSAT
Time Frame: 4 months
Measure: Number; unit: micrograms per deciliter
Arm/Group | All Patients in Study
Number analyzed (Participants) | 1
micrograms per deciliter | 6.2

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=1)
Viral Infection (Infections and infestations) | 1 (1)
Halitosis (Gastrointestinal disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated after one patient was enrolled. Patient discontinued due to lack of improvement in hemoglobin levels and subject compliance issues. Termination after only one subject enrolled does not allow definitive conclusions to be reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT02905981/Prot_SAP_000.pdf